CLINICAL TRIAL: NCT06122506
Title: Nordic Randomized Trial on Laparoscopic Versus Vaginal Cerclage
Acronym: NORACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rigshospitalet, Denmark (Other); Viborg Regional Hospital (Other); Gødstrup Hospital (Other); Aalborg University Hospital (Other); Randers Regional Hospital (Other); Regionshospital Nordjylland (Other Government); Odense University Hospital (Other); Hvidovre University Hospital (Other); Oslo University Hospital (Other); Herlev Hospital (Other); Aarhus University Hospital (Other); Horsens Hospital (Other); Bornholm Hospital, Denmark (Unknown); Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06190; NNF21OC0071037 (Other Grant/Funding Number: Novo Nordic Foundation)
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-09

CONDITIONS: Preterm Birth; Cervical Insufficiency
Keywords: cerclage
MeSH Terms: conditions — Premature Birth; Uterine Cervical Incompetence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Laparoscopic cerclage
  Interventions: Procedure: Laparoscopic cerclage
- Control (Experimental): Vaginal cerclage
  Interventions: Procedure: Vaginal cerclage

INTERVENTIONS:
Procedure: Laparoscopic cerclage — Classic or robot-assisted laparoscopic cerclage in non-pregnant or early pregnant women.
  Other Names: Abdominal cerclage
  Arms: Intervention
Procedure: Vaginal cerclage — Transvaginal cerclage in pregnant women.
  Arms: Control

SUMMARY:
Every year 15 million babies are born prematurely, which can lead to death or life-long disabilities. It is often caused by a dysfunction of the uterine cervix, which constitutes the narrow channel between the vagina and womb. During pregnancy, this channel must remain closed until the beginning of term labor. A weak cervix may not withstand the weight of the fetus, the amniotic fluid and the placenta and the cervical canal will open and cause late miscarriage or preterm delivery. To prevent this, a band (cerclage) can be applied around the cervix either vaginally or laparoscopically prior to a new pregnancy.

To evaluate which treatment is best for most women, we will randomize (allocate by chance) women at risk for preterm birth, to either vaginal cerclage or laparoscopic cerclage in the Nordic countries and England

DETAILED DESCRIPTION:
Both vaginal and abdominal cerclages are procedures that have been used to prevent preterm birth for more than 50 years. However, only one previous study (MAVRIC, Shennan et al. 2020) has compared the two methods in a randomised trial. Other than evidence from the MAVRIC trial there is uncertainty whether an abdominal cerclage should be preferred over vaginal cerclage, and which women would benefit from it the most.

NORACT is an open, multicenter, superiority, randomized controlled trial with the overall objective to compare laparoscopic versus vaginal cerclage in woman in whom the clinician has equipoise as to whether an elective vaginal or abdominal cerclage will be the best intervention to prevent preterm birth. Participants will be recruited pre-pregnancy or in early pregnancy and randomised to vaginal or laparoscopic cerclage. If randomised to laparoscopic cerclage this will be inserted pre-pregnancy or before 10+0 weeks of gestation. The vaginal cerclage will be inserted during pregnancy, before 16+0 weeks of gestation. A total sample of 188 participants will be included to detect a target difference of 15% in the primary outcome between the two groups. The two primary outcomes are delivery before 32+0 weeks of gestation and baby death. The study extends from sites in Denmark, Sweden, Norway, Finland, Iceland, and the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Women in whom the clinician has equipoise as to whether an elective vaginal or abdominal cerclage will be the best intervention to prevent preterm birth.
* Not yet pregnant or <10 weeks' pregnant.

Exclusion Criteria:

* Any circumstance under which the clinician is not willing to randomize is an exclusion criterion.
* Any condition or circumstance under which laparoscopic or vaginal cerclage surgery is contraindicated (i.e. on-going pregnancy of more than 10+0 gestational weeks).
* Language difficulties.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility based on biologic sex.
Enrollment: 188 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Delivery <32+0 weeks of gestation. | At birth.
  In the first subsequent viable pregnancy beyond 14+0 weeks of gestation. First prioritized primary outcome.
Baby death. | From birth - four weeks after due date. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
  Loss of a viable pregnancy beyond 14+0 weeks of gestation, miscarriage, stillbirth or death of a live born infant. Second prioritized primary outcome.

SECONDARY OUTCOMES:
Maternal mortality - surgery related. | 30 days after insertion of laparoscopic or vaginal cerclage.
  Death.
Maternal mortality. | From time of randomisation - 42 days after delivery.
  Death.
Maternal morbidity - surgery related. | 30 days after insertion of laparoscopic or vaginal cerclage.
  Admission to ICU or a unit that provides 24-h medical supervision and is able to provide mechanical ventilation or continuous vasoactive drug support.
Maternal morbidity | From time of randomisation - 42 days after delivery.
  Admission to ICU or a unit that provides 24-h medical supervision and is able to provide mechanical ventilation or continuous vasoactive drug support.
Harm to participant - surgery related. | 30 days after insertion of laparoscopic or vaginal cerclage.
  One or more of the following: Damage to internal organs, need for re-operation, thromboembolic events (defined as deep vein thrombosis, pulmonary embolism or stroke), maternal cardiopulmonary arrest.
Harm to participant | From time of cerclage procedure - 42 days after delivery.
  One or more of the following: Damage to internal organs, thromboembolic events (defined as deep vein thrombosis, pulmonary embolism or stroke), maternal cardiopulmonary arrest.
Bleeding - surgery related. | 30 days after insertion of laparoscopic or vaginal cerclage.
  Blood loss > 500 ml.
Bleeding - pregnancy related. | From time of cerclage procedure - 42 days after delivery.
  Blood loss > 1000 ml.
Maternal infection - surgery related. | 30 days after insertion of laparoscopic or vaginal cerclage.
  Leading to antibiotic treatment, but not ICU.
Maternal infection - pregnancy related. | From time of cerclage procedure - 42 days after delivery
  Leading to antibiotic treatment, but not ICU
Maternal serious infection - pregnancy related. | From time of cerclage procedure - 42 days after delivery.
  Admission to ICU due to serious infection.
Maternal serious infection - surgery related. | 30 days after insertion of laparoscopic or vaginal cerclage.
  Admission to ICU due to serious infection.
PPROM. | At birth.
  Preterm prelabour rupture of membranes, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Threatened preterm labour. | At birth.
  Threatened preterm labour requiring admission and intervention, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Onset of labour. | At birth.
  Spontaneous labor contractions, PROM, induction of labor, c-section. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Mode of birth. | At birth.
  Unassisted vaginal, assisted vaginal (ventouse or forceps), caesarean section (planned, non-planned). In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Modified neonatal mortality. | From birth - four weeks after due date. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
  Death of a liveborn child > 22+0 weeks of gestation.
Neonatal mortality. | From birth - 28 days post delivery. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
  Death in the 1st 28 days of life > 22+0 weeks of gestation.
Fetal loss. | At due date.
  Composite of late miscarriage and stillbirth, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Late miscarriage. | At due date.
  Loss of viable pregnancy between gestational age 14+0-21+6, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Gestational age at birth. | At birth.
  Gestational age at birth, weeks and days, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Delivery < 28 weeks. | At birth.
  Birth before gestational age 28+0, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Delivery < 34 weeks. | At birth.
  Birth before gestational age 34+0, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Delivery < 37 weeks. | At birth.
  Birth before gestational age 37+0, in the first subsequent viable pregnancy beyond 14 weeks of gestation.
Birthweight. | At birth.
  Grams. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Neonatal admission. | From birth - four weeks after due date.
  Number of consecutive days in hospital within 28 days from time of delivery. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
  Any admission counts (SCBU, maternity ward, NICU)
CNS morbidity. | From birth - four weeks after due date.
  Intraventricular Hemorrhage Grade III and IV and/or Periventricular leukomalacia. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Ocular morbidity. | From birth - four weeks after due date.
  Retinopathy requiring treatment. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Gastrointestinal morbidity. | From birth - four weeks after due date.
  Necrotizing Enterocolitis (NEC) and/or SIP (Spontaneous intestinal perforation), requiring surgery. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Respiratory support. | From birth - four weeks after due date.
  Mechanical ventilation or non-invasive ventilation. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Respiratory distress syndrome (RDS). | First two days of life.
  Need for surfactant treatment. In the first subsequent viable pregnancy beyond 14 weeks of gestation.
Early onset neonatal infection. | From birth - four weeks after due date.
  >5 days of i.v. antibiotics, where the treatment commences within the first week of life. In the first subsequent viable pregnancy beyond 14 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Uldbjerg, DMSc, Study Director — Aarhus University Hospital; Julie Glavind, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
After publication of the trial results, the final dataset will be publicly available in an anonymized form using i.e. Zenodo open data repository (CERN) or another equivalent database.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning three months and ending three years after the publication of the last trial results.
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee. Interested parties will be able to request the data by contacting the trial sponsor. Authorship of publications emerging from the shared data will follow standard authorship guidelines and will include authors from the NORACT Board depending on the nature of their involvement.

REFERENCES:
- [Derived] Hansen LK, Krogh LQ, Lantto A, Uldbjerg N, Jensen PT, Shennan A, Hald K, Heikinheimo O, Jacobsson B, Hjartardottir H, Karypidis H, Glavind J. Nordic randomised trial on laparoscopic versus vaginal cerclage (NORACT): trial protocol for an international, multicentre, randomised controlled trial. BMJ Open. 2025 Sep 23;15(9):e107093. doi: 10.1136/bmjopen-2025-107093. PMID 40987744
- See also: Trial website — http://www.noract.dk
- Available data/document: Statistical Analysis Plan — https://drive.google.com/file/d/16iZkdhVtT_pnExSoUhJV5iprYyA1JYhx/view?usp=sharing
- Available data/document: Study Protocol — https://drive.google.com/file/d/1Z_nDas-Emj7x3OnbkcmRl3Pujy0tjlmM/view?usp=sharing